CLINICAL TRIAL: NCT07068100
Title: The Effect of Change Stage-Based Physical Activity Counseling on Physically Inactive Individuals With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ulaş Ar, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-24-6192
Record Dates: First submitted 2024-11-21; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Physical Activity; Behavior Change
Keywords: hypertansion; physical activity; behavior change
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Exercise; Mental Health

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage-of-change based approach to behavior change (Experimental): Participants in the first group will have an individual physical activity program created within the scope of physical activity counseling on the first evaluation day. A 20-30 minute phone call will be made once a week by a psychologist regarding the stage of change they are in, and a 10-15 minute phone call will be made once a week by a physiotherapist for physical activity counseling.
  Interventions: Behavioral: Stage-of-change based physical activity counseling
- Behavior change with brochure (Active Comparator): The second group will be given a brochure with recommendations regarding physical activity and the benefits of physical activity for psychological health.
  Interventions: Behavioral: Giving the group a brochure with recommendations for physical activity and the benefits of physical activity for psychological health

INTERVENTIONS:
Behavioral: Stage-of-change based physical activity counseling — On the first evaluation day, an individual physical activity program will be created for the participants in the group within the scope of physical activity counseling. A 20-30 minute phone call will be made once a week by a psychologist regarding the stage of change they are in, and a 10-15 minute phone call will be made once a week by a physiotherapist for physical activity counseling.
  Arms: Stage-of-change based approach to behavior change
Behavioral: Giving the group a brochure with recommendations for physical activity and the benefits of physical activity for psychological health — The second group will be given a brochure with recommendations for physical activity and the benefits of physical activity for psychological health.
  Arms: Behavior change with brochure

SUMMARY:
Hypertension (HT) is the second most common disease in Turkey and its prevalence is between 30-35%. Adopting healthy lifestyle behaviors can contribute to the prevention of chronic diseases by preserving well-being. However, it has been determined that the control and protection behaviors of HT patients are inadequate. Guidelines for preventing HT recommend weight loss, healthy nutrition, increased physical activity and reduced alcohol consumption. Obesity and lifestyle changes can reduce blood pressure by 5 mmHg. Practices such as not smoking, physical activity (150 minutes per week), Mediterranean diet and alcohol restriction reduce the risk of HT by 50%.

The World Health Organization emphasizes that regular physical activity is important in preventing death and disability. In a study in Turkey involving 15,468 adults, it was determined that only 3.5% of them do regular physical activity. According to the National Household Survey, 20.32% of individuals are sedentary and 15.99% do insufficient physical activity.

Despite the abundance of information on the health benefits of physical activity, the question of why adults do not engage in enough physical activity is important. Research is insufficient for physical activity knowledge and behavior change in individuals. Physical activity increase interventions based on theories such as the Transtheoretical Model (TM) are effective for behavior change. TM includes elements such as stages of change, self-efficacy, and decision-making balance.

The aim of this study was to investigate the effects of individual physical activity counseling based on the stage of change in physically inactive hypertensive individuals on physical activity levels and the perceived benefits and barriers of individuals' participation in physical activity.

DETAILED DESCRIPTION:
Hypertension (HT) is the second most commonly diagnosed condition in Turkey and represents a global health issue. Studies indicate that the prevalence of HT in Turkey ranges from 30% to 35%, with a steadily increasing trend. When healthy lifestyle behaviors become ingrained attitudes, they can contribute to maintaining well-being and improving health status, thereby preventing chronic diseases. However, patients' attitudes and behaviors regarding HT management and preventive measures have been found to be inadequate. Guidelines for HT prevention target modifiable risk behaviors such as weight loss, healthy eating, increased physical activity, and reduced alcohol consumption. Changes that can positively impact blood pressure include increased physical activity, reduced salt intake, smoking cessation, weight loss, alcohol restriction, and the adoption of a healthy dietary pattern.

In 2013, the American Heart Association, the American Hypertension Association, and the European Hypertension Association published lifestyle modification recommendations consistent with the Dietary Approaches to Stop Hypertension (DASH), emphasizing a sodium intake of less than 1.5-2.3 grams per day, weight loss for individuals with a body mass index (BMI) >25, alcohol intake limited to 10-20 grams per day, and aerobic exercise targeting 150 minutes per week. Each of these interventions is expected to reduce systolic blood pressure (SBP) by 4-6 mmHg in a dose-dependent and additive manner. Addressing factors contributing to HT etiology, such as obesity, dietary excesses (high sodium, inadequate potassium, calcium, magnesium, protein, fiber, and omega-3 fatty acids), alcohol consumption, and physical inactivity, can collectively reduce blood pressure by an average of 5 mmHg. In the SUN cohort, adherence to non-smoking, physical activity (150 minutes/week), a Mediterranean diet, and maintaining a BMI of less than 22 in men and 25 in women, along with either abstaining from or limiting alcohol consumption, was associated with nearly a 50% reduction in HT risk. Smoking has been noted to increase SBP by 4 mmHg compared to placebo.

In recent years, the importance of reducing sedentary lifestyles and increasing physical activity for public health has gained recognition. There is substantial evidence of the numerous physiological and psychological benefits of physical activity, including the prevention or improvement of coronary heart disease, hypertension, type II diabetes, colon cancer, obesity, stress, and depression. Physical activity is defined as any bodily movement produced by skeletal muscles that require energy expenditure, encompassing not only sports activities but also exercise, household chores, and workplace physical activities.

Data from the World Health Organization (WHO) indicate that physical inactivity is among the top ten global causes of mortality and disability. WHO recommends that regular moderate-intensity physical activity be performed for at least 30 minutes on most days of the week. However, 60-85% of the global population does not engage in the recommended level of physical activity. In a 2004 study conducted by the Turkish Ministry of Health titled "Healthy Eating, Protecting Our Hearts," physical activity habits were surveyed among 15,468 adults from seven provinces, revealing that only 3.5% engaged in regular physical activity (defined as at least three days per week of moderate intensity for 30 minutes). According to the National Household Research (2006), 20.32% of individuals over 18 years of age in Turkey were found to be sedentary, and 15.99% exhibited insufficient levels of physical activity.

Despite extensive knowledge regarding the health benefits of physical activity, many adults do not engage in sufficient physical activity. Research suggests that mere knowledge about physical activity is insufficient for behavior change. Robbins et al. indicated that lifelong physical activity can be promoted through theory-based interventions. Studies have shown that interventions aimed at increasing physical activity grounded in the Transtheoretical Model (TM) are effective. Developed by Prochaska and DiClemente in 1982, TM is a promising internationally recognized model for health behavior change, comprising four elements: stages of change, self-efficacy, decisional balance, and processes of change. The stages of change define the time dimension of behavior modification, explaining the timing of individuals' intentions, attitudes, and behavior changes. Progress through these stages also signifies an individual's readiness to engage in regular physical activity. The physical activity behavior change process consists of five stages: pre-contemplation, contemplation, preparation, action, and maintenance.

The Theory of Planned Behavior (TPB), developed by Ajzen in 1985, is one of the most widely used theories to explain human behavior and is applied in physical activity research. In TPB, the key factor is the individual's intention to perform a specific behavior; thus, measuring intention is critical for behavior change. Research findings support the use of the Theory of Planned Behavior in measuring physical activity intentions and predicting behavior.

This study aims to investigate the effects of stage-based individual physical activity counseling on the physical activity levels of physically inactive individuals with hypertension, as well as to explore the perceived benefits and barriers to participation in physical activity among these individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-60
2. Not doing a minimum of 150 minutes/week of moderate intensity or 75 minutes/week of vigorous intensity physical activity
3. Being willing to participate in the study,
4. Not having problems reading and/or understanding the scales and being able to cooperate with the tests,
5. Having stable and controlled hypertension.

Exclusion Criteria:

1. Active infection,
2. Having a musculoskeletal or neurological disease that may affect exercise performance, symptomatic heart disease,
3. Having a neurological disease or other clinical diagnosis that may affect cognitive status,
4. Having any orthopedic or neuromuscular disorder that will prevent walking or exercise performance,
5. Having any chronic disease or having psychiatric disorders or mental disorders that may prevent cooperation.
6. Being in the maintenance phase according to the change phase diagnosis form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity | through study completion, an average of 1 year
  The long form of the International Physical Activity Questionnaire (IPAQ) will be used. The International Physical Activity Questionnaire - Long Form (IPAQ-LF) is a validated tool used to assess an individual's physical activity across various domains, including work, transport, domestic, and leisure-time activities. Physical activity levels are expressed in MET-minutes per week, where MET stands for Metabolic Equivalent of Task-a unit that estimates the energy expenditure of physical activities. One MET is defined as the energy cost of sitting quietly, equivalent to approximately 3.5 mL of oxygen consumption per kg of body weight per minute. Based on IPAQ scoring guidelines, total physical activity can range from a minimum of 0 MET-min/week (no reported activity) to a maximum of over 20,000 MET-min/week or more in highly active individuals. In this study, IPAQ-LF will be used to quantify participants' physical activity levels and categorize them as low, moderate, or high activity.
Behavior Change | through study completion, an average of 1 year
  The Stage of Change Identification Form will be used to determine the stage of behavioral change that individuals are in.

SECONDARY OUTCOMES:
Comorbidity | through study completion, an average of 1 year
  The Charlson Comorbidity Index (CCI) is a validated tool used to predict mortality risk by quantifying the burden of comorbid conditions. It assigns weighted scores to 17 different chronic diseases based on their severity and prognostic impact. Conditions such as myocardial infarction, diabetes, chronic pulmonary disease, and malignancy are scored from 1 to 6 points. The total CCI score is calculated by summing these weights, with a minimum score of 0 (no comorbidities) and no fixed maximum, though scores typically range up to 33 in clinical populations. Higher CCI scores indicate greater comorbidity burden and are associated with increased risk of mortality.
Self care | through study completion, an average of 1 year
  The Hypertension Self-Care Profile - High Blood Pressure Inventory (Version 3) is a psychometric tool designed to assess self-care behaviors in individuals with hypertension. It evaluates key domains such as medication adherence, diet, physical activity, blood pressure monitoring, weight management, and alcohol and tobacco use. Items are rated using a Likert scale, and total scores reflect the level of engagement in self-care practices, with higher scores indicating better self-care behavior. The total score typically ranges from 0 to 180, depending on the version and number of items used. In this study, this inventory will be used to evaluate participants' self-care capacity and adherence to hypertension management recommendations.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diaz-Gutierrez J, Ruiz-Estigarribia L, Bes-Rastrollo M, Ruiz-Canela M, Martin-Moreno JM, Martinez-Gonzalez MA. The role of lifestyle behaviour on the risk of hypertension in the SUN cohort: The hypertension preventive score. Prev Med. 2019 Jun;123:171-178. doi: 10.1016/j.ypmed.2019.03.026. Epub 2019 Mar 19. PMID 30902699